CLINICAL TRIAL: NCT03960788
Title: Gadoxetate Sodium Enhanced Magnetic Resonance Imaging (MRI) as a Biomarker for Aggressive Prostate Cancer
Brief Title: Gadoxetate Sodium Enhanced MRI as a Biomarker for Aggressive Prostate Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sadhna Verma, Adjunct Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EOVIST
Record Dates: First submitted 2019-04-23; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cancer of the Prostate; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRI with Gadoxetate Sodium (Experimental): Subjects will receive Gadoxetate Sodium during MRI.
  Interventions: Drug: Gadoxetate Sodium

INTERVENTIONS:
Drug: Gadoxetate Sodium — Gadoxetate Sodium is an FDA approved contrast agent to be used during magnetic resonance imaging.

SUMMARY:
The purpose of this research study is to test to see if Gadoxetate Sodium is a useful contrast agent for detecting prostate cancer during magnetic resonance imaging (MRI). Gadoxetate Sodium is an FDA approved contrast agent that is currently used to detect liver cancer. Gadoxetate Sodium shows promise in identifying more aggressive prostate cancers at earlier stages. The study will also test to see if specific genes are expressed in the left over tissue samples from previous prostate fusion biopsy. The investigators hypothesize that Gadoxetate Sodium-enhanced MRI can differentiate aggressive prostate cancer and predict its early recurrence.

DETAILED DESCRIPTION:
A substantial body of evidence implicates androgen hormones, such as testosterone, play a key role in aggressive prostate carcinogenesis, and much work has been done to evaluate the relationship between the concentration of testosterone and clinical outcome of patients with prostate cancer. Several uptake transporters localized to the cell membrane have shown to enhance steroid hormone uptake, and these same transporters are also expressed within the prostate where they could increase the capability of neoplastic cells to use testosterone. One group of uptake carriers is the organic anion-transporting polypeptide (OATP) superfamily encoded by SLCO genes. OATPs are localized to normal human hepatocytes. OATP1B3, a member of this family, is also expressed by cancer cells derived from aggressive prostate cancer. Studies have shown that in prostate cancer, testosterone uptake by cells occurs via OATP1B3, and its presence increases from undetectable levels in normal prostatic tissue and benign hyperplasia to marked expression in aggressive prostate cancer.

Current prostate cancer (PCa) diagnosis methods have false positives and are limited in predicting cancer recurrence. Gadoxetate Sodium is a magnetic resonance imaging agent which is FDA-approved gadolinium chelate for detecting hepatocellular carcinoma, as normal hepatocytes express OATP1B3 while most hepatocellular carcinomas do not. Gadoxetate Sodium acts as a substrate for OTAP1B3, therefore, OATP1B3 positive prostate tumors can potentially be visualized on MR imaging. Making this contrast agent useful in the evaluation of OATP1B3 status in patients with aggressive PCa and potentially serve as a prognostic and treatment biomarker.

The investigators hypothesize that Gadoxetate Sodium -enhanced MRI can differentiate aggressive PCa and predict its early recurrence. The investigators aim to enroll 50 patients and sort them into localized or metastatic PCa, based on tumor grade. Subjects that agree to participate will be scheduled for a research pelvic MRI with the Gadoxetate Sodium contrast within 3 weeks of their office visit. The procedure is be conducted as a standard pelvic MRI but instead of gadolinium contrast being administered, Gadoextate Sodium will be dosed at 0.1/mL per kilogram of body weight (as prescribed on the contrast label). Once the subject has undergone the research MRI scan using Gadoxetate Sodium, the MRI and assigned enhancement ratios will be reviewed. Contrast enhancement ratios (CERs) will be calculated to evaluate the difference in the degree of enhancement between the tumors and normal tissue. Subject demographic information, medical history and enhancement ratios will be recorded in the study database.

Previously obtained remnant biopsy samples from enrolled subjects will be used for transcriptome and epigenome profiling using genome-wide and targeted gene approaches.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 18 years old.
* Subjects with clinically localized OR advanced prostate cancer with biopsy confirmation and sufficient tissue available (obtained before Gadoxetate Sodium injection) for OATP1B3 expression.
* Subjects must have a prior MRI with gadolinium obtained as part of their standard of care for comparison available. This may have been obtained as part of an image guided biopsy.
* Serum creatinine within 3 weeks prior to Gadoxetate Sodium MRI less than or equal to 1.8mg/dl and estimated glomerular filtration rate (eGFR) must be greater than 60 ml/min/1.73m.
* Patients must have normal liver function as defined below: total bilirubin less than 2 times normal institutional limits or greater than 3.0 mg/dl in patients with Gilbert s syndrome AST(SGOT) and ALT(SGPT) less than or equal to 3 times institutional upper limit of normal
* Ability of subject to sign a written informed consent document.

Exclusion Criteria:

* Subjects that have received a prostatectomy
* Subjects with known hypersensitivity and allergy to gadolinium contrast agents
* Subjects with chronic kidney disease or acute kidney injury. Chronic Kidney disease is GFR<30. Acute kidney injury (AKI) is defined as an abrupt or rapid decline in renal filtration function and is screened by excluding patient's that have a GFR <60 within 3 weeks of their scan, as well as screening patients on the day of the scan for kidney disease and contraindications using the standard form based on the Updated ACR Screening Recommendations on Gadolinium Based MR Contrast Agents, Renal Disease Patients. Patients who show signs of renal disease from this form will be excluded from the study.
* Subjects with contraindications to MRI
* Subjects with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Males may apply due to condition under study.
Enrollment: 50 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of Gadoxetate Sodium to gadolinium in effectiveness of identification of prostate cancer as measured by contrast enhancement ratios | 3 weeks from consent
  This single outcome will be measured by comparing the contrast enhancement ratio from pre-study images from participating subjects originally imaged with gadolinium enhanced contrast against contrast enhancement ratios from subjects receiving Gadoxetate Sodium enhanced scans. The measurements taken using the enhancement ratios will be for two areas of interest in the prostate in tumor tissue and these will be collected from pre-study, and post-study images only.
  A contrast enhancement ratio is a quantitative measure used to assess the degree of enhancement (brightness) between normal and abnormal tissue in imaging.

SECONDARY OUTCOMES:
Comparison of the contrast enhancement ratio of OATP1B3 + and - samples taken from post-Gadoxetate Sodium subjects to determine if Gadoxetate Sodium to determine if it differentiates androgen resistant cancers. | 3 weeks from consent
  This single outcome will be measured by collecting a tumor tissue biopsy post scan with Gadoxetate Sodium, performing a molecular analysis for the genetic marker OATP1B3 (agent present in resistant cancers) and comparing the contrast enhancement ratio in those samples that have OATP1B3 to those samples without.
  A contrast enhancement ratio is a quantitative measure used to assess the degree of enhancement (brightness) between normal and abnormal tissue in imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Sadhna Verma, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No